CLINICAL TRIAL: NCT00790179
Title: Continuous Lumbar Plexus Block for Postoperative Pain Control After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Joseph Marino M.D., Huntington Hospital, North Shore-LIJ Health System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1989md
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Postoperative Pain
Keywords: Continuous lumbar plexus,Femoral,hydromorphone
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PCA;active comparator (Active Comparator): Patients with intravenous PCA hydromorphone alone
  Interventions: Procedure: continuous infusion of ropivacaine via CLPB vs. CFB vs IV PCA
- CFB (Active Comparator): Patients with a continuous femoral block (CFB) + PCA hydromorphone
  Interventions: Procedure: continuous infusion of ropivacaine via CLPB vs. CFB vs IV PCA
- CLPB (Active Comparator): Patients with a continuous lumbar plexus block + PCA hydromorphone
  Interventions: Procedure: continuous infusion of ropivacaine via CLPB vs. CFB vs IV PCA

INTERVENTIONS:
Procedure: continuous infusion of ropivacaine via CLPB vs. CFB vs IV PCA — 0.5% Ropivacaine bolus of 30 ml. followed by ropivacaine 0.2%at 10 ml/hr via CLPB vs. CFB.
  Hydromorphone 0.3 mg demand only every 10 minutes via IV PCA.

SUMMARY:
Continuous lumbar plexus and femoral blocks have been demonstrated to provide effective postoperative analgesia of the lower extremity following total joint arthroplasty. The purpose of this study was to compare these two techniques when used with intravenous patient-controlled analgesia and the use of patient-controlled analgesia alone for postoperative pain management following unilateral total hip arthroplasty.

DETAILED DESCRIPTION:
above may be applied

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* primary diagnosis of osteoarthritis

Exclusion Criteria:

* allergy to local anesthetics
* peripheral neuropathy
* opioid dependency
* dementia
* coagulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2003-01; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
VAS pain scores | at 24 and 48 hours

SECONDARY OUTCOMES:
hydromorphone consumption,patient satisfaction,distance ambulated, opioid-related side effects | at 24 and 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Marino, M.D., Principal Investigator — Huntington Hospital